CLINICAL TRIAL: NCT05967260
Title: A Crossover Study to Assess the Effect of an Artificial Intelligence (AI)-Based Bedtime Smart Snack Intervention in Preventing Overnight Low Glucose in People With T1D on Multiple Daily Injections.
Brief Title: DailyDose Smart Snack Study for T1D on MDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Clara Mosquera-Lopez, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25174
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia
Keywords: Decision Support; Dexcom CGM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Participants will use the DailyDose Smart Snack smart phone application which contains an AI-based model that predicts the likelihood of overnight low glucose at bedtime every night and will recommend a personalized snack to help avoid nocturnal hypoglycemia. The nutritional content of the snack (carbohydrate, protein, fat, etc.) will be dependent on the predicted overnight minimum glucose and the predicted time of the minimum overnight glucose level. During this arm, participants will also be asked to wear a smart watch overnight, weigh themselves weekly, and answer a one-item sleep quality scale survey weekly.
  Interventions: Device: DailyDose Smart Snack app
- Control (Active Comparator): Participants will wear Dexcom G6 CGM and will manage their glucose as usual. Participants will be asked to wear a smart watch overnight to collect sleep metrics, weigh themselves weekly in the morning before eating, and answer a one-item sleep quality scale survey weekly.
  Interventions: Device: Dexcom G6 CGM

INTERVENTIONS:
Device: DailyDose Smart Snack app — A decision support tool that predicts the likelihood of overnight low blood sugar based on current CGM and inputted exercise. App will recommend a snack at bedtime based on the minimum low glucose predicted and the time of the low glucose.
  Arms: Intervention
Device: Dexcom G6 CGM — A commercially available Continuous Glucose Monitoring system that utilizes a transmitter and sensor to measure sensor glucose levels that transmit to a smart phone app.
  Arms: Control

SUMMARY:
This is a single-center, open-label, crossover trial with two arms and two periods (2x2) and one-week washout period. The study is designed to evaluate the efficacy of an AI-based bedtime smart snack intervention in reducing nocturnal low glucose in people living with T1D on MDI therapy compared with traditional CGM-augmented MDI therapy as the control.

DETAILED DESCRIPTION:
Participants will be randomized to either first use CGM only to manage glucose for four weeks (control arm) followed by four weeks of DailyDose App + bedtime smart snack intervention (intervention arm), or vice-versa. There will be a one-week washout period between arms.

During the control arm, participants will wear CGM and will manage their glucose as usual. Participants will be asked to wear a smart watch overnight to collect sleep metrics, weigh themselves weekly in the morning before eating, and answer a one-item sleep quality scale survey weekly. We will collect CGM measurements during the control arm for evaluation of effect of intervention and assessment of the accuracy of low glucose prediction.

During the intervention arm, participants will use the DailyDose Smart Snack smart phone app. When they are getting ready for bed, an AI-based model in DailyDose will predict the likelihood of overnight low glucose at bedtime and will recommend a personalized snack to help avoid nocturnal hypoglycemia. The nutritional content of the snack (carbohydrate, protein, fat, etc.) will be dependent on the predicted overnight minimum glucose and the predicted time of the minimum overnight glucose level. During this arm, participants will also be asked to wear a smart watch overnight, weigh themselves weekly, and answer a one-item sleep quality scale survey weekly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year
* Male or female participants 18 years of age or older
* Using multiple daily injections
* HbA1c <10% at screening
* Current use of a continuous glucose monitoring system with at least two episodes of overnight hypoglycemia (defined as sensed glucose <70 mg/dL for at least 10 minutes between the hours of 10 PM and 6 AM) within 30 days prior to screening
* Individuals with history of severe hypoglycemia requiring third party assistance must have a companion in the same dwelling as the study participant who will be linked to the participant's Dexcom app during the control arm of the study, and who is trained in the administration of glucagon.
* Willingness to follow all study procedures
* Willingness to sign informed consent and HIPAA documents

Exclusion Criteria:

* Individual of childbearing potential who is pregnant or intending to become pregnant or breast-feeding or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide, and the man uses a condom), or abstinence
* Any active infection
* Known or suspected abuse of alcohol, narcotics, or illicit drugs (except marijuana use)
* Seizure disorder
* Use of non-insulin glucose lowering medications
* Use of steroids
* Stage-three or more advanced chronic kidney disease
* Hypo- or hyper- thyroidism that is not medically optimized and on a stable regimen define as Thyroid-stimulating hormone (TSH) outside of the normal reference range based on screening labs
* Adrenal insufficiency
* Cirrhosis
* Any life-threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the participant's safety or compliance with the protocol
* Individual working night shifts

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control to Intervention: The randomization order for participants in this arm was Dexcom G6 CGM (control) followed by DailyDose Smart Snack (intervention). Each arm was 4 weeks long.
- Intervention to Control: The randomization order for participants in this arm was DailyDose Smart Snack (intervention) followed by Dexcom G6 CGM (control). Each arm was 4 weeks long.
Period: First Rest Period (1-12 Weeks)
Arm/Group | Control to Intervention | Intervention to Control
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Period: First Arm Start-up Visit (4 Weeks)
Arm/Group | Control to Intervention | Intervention to Control
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Dexcom CGM failed while participant out of town without ability to receive a replacement | 0 | 1
Period: Second Rest Period (1-4 Weeks)
Arm/Group | Control to Intervention | Intervention to Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Arm Start-up Visit
Arm/Group | Control to Intervention | Intervention to Control
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Period: Third Rest Period (1-2 Weeks)
Arm/Group | Control to Intervention | Intervention to Control
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Study Completion Visit
Arm/Group | Control to Intervention | Intervention to Control
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control to Intervention | Intervention to Control | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (14.6) | 37 (15.1) | 39 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 7 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Probability of Overnight Hypoglycemia
Description: An episode of overnight hypoglycemia is counted if sensor glucose is <70 mg/dL for at least two measurements during an eight-hour period following announced bedtime. This is assessed by number of episodes divided by total number of nights.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of nights
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of nights | 23.6 (15.6) | 26.0 (14.1)

2. Secondary Outcome: Time to the First Overnight Low-glucose Event (<70 mg/dL)
Description: Number of hours until first CGM measurement <70 mg/dL when CGM remains < 70 mg/dL for at least 10 minutes.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
hours | 2.8 (1.4) | 3.3 (1.4)

3. Secondary Outcome: Percentage of Time With Sensed Glucose Less Than 54 mg/dL (Overnight)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are less than 54 mg/dL overnight (announced bedtime + 8 hours).
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 1.0 (1.5) | 1.3 (3.2)

4. Secondary Outcome: Percentage of Time With Sensed Glucose Less Than 54 mg/dL (24-hour/Day Study Duration)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are less than 54 mg/dL across the full 24-hour/day study duration.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 0.7 (0.7) | 0.7 (1.0)

5. Secondary Outcome: Percentage of Time With Sensed Glucose Less Than 70 mg/dL (Overnight)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are less than 70 mg/dL overnight (announced bedtime + 8 hours).
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 4.2 (3.8) | 4.7 (5.5)

6. Secondary Outcome: Percentage of Time With Sensed Glucose Less Than 70 mg/dL (24-hour/Day Study Duration)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are less than 70 mg/dL across the 24-hour/day study duration.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 3.2 (1.8) | 3.1 (2.3)

7. Secondary Outcome: Percentage of Time With Sensed Glucose Between 70-180 mg/dL (Overnight)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are between 70 and 180 mg/dL overnight (announced bedtime + 8 hours).
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 64.0 (14.4) | 61.8 (14.8)

8. Secondary Outcome: Percentage of Time With Sensed Glucose Between 70-180 mg/dL (24-hour/Day Study Duration)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are between 70 and 180 mg/dL across the full 24-hour/day study duration.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 63.9 (14.9) | 61.4 (16.5)

9. Secondary Outcome: Percentage of Time With Sensed Glucose Greater Than 180 mg/dL (Overnight)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are greater than 180 mg/dL overnight (announced bedtime + 8 hours).
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 31.7 (15.6) | 33.5 (16.1)

10. Secondary Outcome: Percentage of Time With Sensed Glucose Greater Than 180 mg/dL (24-hour/Day Study Duration)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are greater than 180 mg/dL across the full 24-hour/day study duration.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 32.8 (15.3) | 35.5 (16.6)

11. Secondary Outcome: Percentage of Time Sensed Glucose Greater Than 250 mg/dL (Overnight)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are greater than 250 mg/dL overnight (announced bedtime + 8 hours).
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 10.2 (8.9) | 9.7 (9.0)

12. Secondary Outcome: Percentage of Time Sensed Glucose Greater Than 250 mg/dL (24-hour/Day Study Duration)
Description: Assess the mean percentage of time that the Dexcom G6 reported sensor glucose values are greater than 250 mg/dL across the full 24-hour/day study duration.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
percentage of time | 10.4 (9.5) | 11.3 (10.8)

13. Secondary Outcome: Mean Sensed Glucose (Overnight)
Description: Assess the mean reported sensor glucose values overnight (announced bedtime + 8 hours) using the Dexcom sensor.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
mg/dL | 159.0 (25.1) | 160.4 (26.5)

14. Secondary Outcome: Mean Sensed Glucose (24-hour/Day Study Duration)
Description: Assess the mean reported sensor glucose values across the full 24-hour/day study duration using the Dexcom sensor.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
mg/dL | 161.9 (24.2) | 165.2 (27.3)

15. Secondary Outcome: Accuracy of Overnight Low Glucose Prediction by Sensitivity
Description: Assessment of accuracy of the overnight low glucose prediction algorithm by sensitivity. This is measured by the number of true positives that the algorithm predicts hypoglycemia overnight divided by all of the hypoglycemic events.
Time Frame: 4 weeks of control period
Measure: Number; unit: percentage of true positive events
Groups:
- Control Arm: A total of 540 nights across all 20 participants who completed the study had sufficient data to be included in the analysis which assumes the minimum nocturnal glucose would have been <70 mg/dL without AI-detected carbohydrate. intake
Arm/Group | Control Arm
Number analyzed (Participants) | 20
percentage of true positive events | 71.6

16. Secondary Outcome: Accuracy of Overnight Low Glucose Prediction by Specificity
Description: Assessment of accuracy of the overnight low glucose prediction algorithm by specificity. This is measured by calculating 1.0 minus the false positive rate for overnight hypoglycemia prediction.
Time Frame: 4 weeks of control period
Measure: Number; unit: percentage of true negative events
Arm/Group | Control Arm
Number analyzed (Participants) | 20
percentage of true negative events | 56.8

17. Secondary Outcome: Change in Weight
Description: Asses mean weight change from start to end of each arm.
Time Frame: 8 weeks (4-week control period vs. 4-week intervention period)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
kg | -2.1 (3.0) | -0.7 (1.3)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: All participants that began/started the first rest period after randomization are included in the adverse events. The numbers from the participant flow indicate that 21 subjects began the first rest period.
Groups:
- Active Comparator: Control: Participants will wear Dexcom G6 CGM and will manage their glucose as usual. Participants will be asked to wear a smart watch overnight to collect sleep metrics, weigh themselves weekly in the morning before eating, and answer a one-item sleep quality scale survey weekly.
- Experimental: Intervention: Participants will use the DailyDose Smart Snack smart phone application which contains an AI-based model that predicts the likelihood of overnight low glucose at bedtime every night and will recommend a personalized snack to help avoid nocturnal hypoglycemia. The nutritional content of the snack (carbohydrate, protein, fat, etc.) will be dependent on the predicted overnight minimum glucose and the predicted time of the minimum overnight glucose level. During this arm, participants will also be asked to wear a smart watch overnight, weigh themselves weekly, and answer a one-item sleep quality scale survey weekly.
Arm/Group | Active Comparator: Control | Experimental: Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Control (N=20) | Experimental: Intervention (N=20)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05967260/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT05967260/ICF_002.pdf